CLINICAL TRIAL: NCT02003157
Title: Efficacy of Hypnosis During Embryo Transfer Procedure on Clinical Pregnancy Rate for Patients Undergoing Assisted Reproductive Technology IVF or ICSI
Acronym: HYPNOART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011 A00081-40
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2011-10

CONDITIONS: Infertility
Keywords: hypnosis embryo transfer IVF ICSI
MeSH Terms: conditions — Infertility

ARMS (2):
- hypnosis (Active Comparator): embryo transfer procedure with hypnosis
  Interventions: Procedure: hypnosis during embryo transfer or usual transfer procedure
- usual (Active Comparator): embryo transfer usual procedure
  Interventions: Procedure: hypnosis during embryo transfer or usual transfer procedure

INTERVENTIONS:
Procedure: hypnosis during embryo transfer or usual transfer procedure

SUMMARY:
The purpose of this study is to compare the clinical benefits that can be expected by the Embryo transfert procedure with hypnosis to the usual embryo transfer procedure

ELIGIBILITY:
Inclusion Criteria:

Consent to participate in study Age ≥ 18 years and < 41 years IVF or IVF/ICSI attempt GnRH antagonist or agonist stimulation protocol Scheduled transfer of 1 or 2 embryos

Exclusion Criteria:

Refusal to provide consent refusal hypnosis FSH > 13 mUImL CFA < 8 follicles AMH < 0.5 ngml Patient not covered by the social security system (NHS)

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | between weeks 5 and 7 after embryo transfer
  sonography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU angers, Angers, Angers, France